CLINICAL TRIAL: NCT05187039
Title: Evaluation of Atelectasis Formation and Regression With Electrical Impedance Tomography in the Perioperative Phase of Obese Patients Scheduled for Laparoscopic Bariatric Surgery
Brief Title: Bariatric Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01473
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia
Keywords: Bariatric; Obese; Laparoscopic; Electrical impedance tomography
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electrical impedance tomography during anesthesia — Thoracic electrical impedance tomography measurements ( min each) will be performed at the following time points: before induction of the anaesthesia; before the surgical procedure when the induction is terminated and recruitment manoeuvers have been performed; after the termination of the surgical procedure; before transport to the Post anaesthesia Care Unit (PACU); before the discharge from the PACU after 2 hours of monitoring. An additional thoracic EIT-measurement will be performed before discharge at home. For this, resulting potential differences are measured, and impedance distribution sampled at 30 Hz will be calculated. Relative change in poorly ventilated lung regions (silent spaces) and end-expiratory lung impedance (EELI) and measures of ventilation inhomogeneity will be calculated using customised code (Matlab R2021a, The MathWorks, Nattick, Massachusetts, USA).

SUMMARY:
This study investigates under controlled conditions the variation of poorly ventilated lung units (silent spaces) in obese patients scheduled for laparoscopic bariatric surgery in the perioperative phase.

DETAILED DESCRIPTION:
Eligible patients with written informed consent, scheduled for laparoscopic bariatric surgery. As for standard of care no premedication will be given for bariatric patients. Patients will be monitored according the local standard.

Thoracic electrical impedance tomography measurements (each measurement will last 1 min) will be performed at the following time points: before induction of the anaesthesia; before the surgical procedure when the induction is terminated and recruitment manoeuvers have been performed; after the termination of the surgical procedure; before transport to the Post anaesthesia Care Unit (PACU); before the discharge from the PACU after 2 hours of monitoring. An additional thoracic electrical impedance tomography measurement (duration 1 min) will be performed before discharge at home. For this, resulting potential differences are measured, and impedance distribution sampled at 30 Hz will be calculated by an automated linearized Newton-Raphson reconstruction algorithm. Relative change in poorly ventilated lung regions (silent spaces) and end-expiratory lung impedance (EELI) and measures of ventilation inhomogeneity such as the global inhomogeneity index will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40
* ASA physical status 1 to 4
* Over 18 years of age providing written informed consent

Exclusion Criteria:

* BMI <40
* Known severe pulmonary hypertension,
* Need of home oxygen therapy
* Known heart failure
* Suspected, or known recent pulmonal infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include obese patients exceeding body mass index (BMI) 40, scheduled for laparoscopic bariatric surgery at the University Hospital - Inselspital in Bern
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Proportion of poorly ventilated lung areas (silent spaces) | 2 hours
  Proportion of poorly ventilated lung areas (silent spaces) by using electrical impedance tomography (EIT) before the discharge from PACU (two hours after admission to PACU).

SECONDARY OUTCOMES:
EIT-Measurement after the end of induction before the surgical procedure | 2 minutes after the end of anesthesia induction
  Detection of changes in silent spaces, ventilation inhomogeneity and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT)
EIT-Measurement at the end of the surgical procedure | 5 minutes after Capnoperitoneum
  Detection of changes in silent spaces, ventilation inhomogeneity and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT)
EIT-Measurement 2 minutes after the end of anaesthesia, before the transport in PACU | 2 minutes after the end of anaesthesia, before the transport to PACU.
  Detection of changes in silent spaces, ventilation inhomogeneity and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT)
EIT-Measurement before discharge from the PACU | Two hours after admission of the patient at PACU, before first mobilisation and before discharge from PACU
  Detection of changes in silent spaces, ventilation inhomogeneity and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT)
EIT-Measurement before discharging the patient at home | At hospital discharge, up to 3 days
  Detection of changes in silent spaces, ventilation inhomogeneity and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT)
Duration of surgical procedure. | Up to 90 to 150 minutes
  Duration of surgical procedure.
Duration of anaesthesia | Up to 90 to 180 minutes
  Duration of anaesthesia
Desaturation below 90%. | During anaesthesia monitoring, from 1 to 10 minutes
  Difference of formation and course of silent lung areas in patients with and without pre-existing CPAP-therapy
Follow up at 14 days | 14 days
  Follow-up by phone, regarding respiratory complications or need for rehospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Braun, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No